CLINICAL TRIAL: NCT02530060
Title: An Open-Label Study to Evaluate the Pharmacokinetics of Rilpivirine/Tenofovir/Emtricitabine After a Single-Oral Administration of a Rilpivirine/Tenofovir Disoproxil Fumarate/Emtricitabine Fixed-Dose Combination Tablet in Healthy Japanese Adult Male Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics of Rilpivirine/Tenofovir/Emtricitabine After a Single-Oral Administration in Healthy Japanese Adult Male Participants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR107748; TMC278FDCHIV4001 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2015-08-19; First posted 2015-08-20 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
Keywords: Healthy; Rilpivirine; Tenofovir; Emtricitabine; Tenofovir Disoproxil Fumarate
MeSH Terms: interventions — Rilpivirine; Emtricitabine, Rilpivirine, Tenofovir Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rilpivirine/Tenofovir Disoproxil Fumarate/Emtricitabine (Experimental): Participants will receive single oral dose of fixed dose combination (FDC) tablet comprising of Rilpivirine/Tenofovir Disoproxil Fumarate/Emtricitabine on Day 1.
  Interventions: Drug: Rilpivirine/Tenofovir Disoproxil Fumarate/Emtricitabine FDC

INTERVENTIONS:
Drug: Rilpivirine/Tenofovir Disoproxil Fumarate/Emtricitabine FDC — Fixed dose combination tablet contains 25 milligram (mg) of Rilpivirine, 300 mg of Tenofovir Disoproxil Fumarate (TDF) and 200 mg of Emtricitabine (FTC).
  Other Names: Complera

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) of rilpivirine/Tenofovir/Emtricitabine (RPV/TFV/FTC) after a single-oral administration of Complera (the fixed-dose combination of RPV, FTC, Tenefovir disoproxil fumarate [TDF]) to healthy Japanese adult male participants.

DETAILED DESCRIPTION:
This is a single center, open-label, single oral dose study in healthy Japanese adult male participants. The study consists of 3 phases; a screening phase up to 27 days (Day -28 to Day -2), an in-patient phase from Day -1 to Day 3 (dosing day is Day 1), and a follow-up assessment phase from Day 4 to the last follow-up assessment scheduled on Day 15 or at the time of early withdrawal. All participants will receive a single oral dose of one Complera tablet on Day 1 within 5 minutes after completion of the standardized breakfast. Pharmacokinetics of RPV/TFV/FTC will be assessed as the primary objective of the study. Safety of each participant will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Willing to adhere to the prohibitions and restrictions specified in this protocol
* Participant who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control eg, either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 3 months after receiving the dose of study drug
* Body mass index (BMI) between 18 and 30 kilogram per meter square (kg/m^2) (inclusive), and body weight not less than 50 kg
* Blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeters of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic
* Non-smoker or participant who habitually smokes no more than 10 cigarettes or equivalent of e-cigarettes, or 2 cigars, or 2 pipes of tobacco per day for at least 6 months before first study drug administration

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency (creatinine clearance below 60 mL/min), thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening or at admission to the study center as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs, or 12 lead electrocardiogram (ECG) at screening or at admission to the study center as deemed appropriate by the investigator
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements) within 14 days before the first dose of the study drug is scheduled until completion of the study
* History of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (4th edition text revision or 5th edition) (DSM-IV or DSM-5) criteria or International Statistical Classification of Diseases and Related Health Problems 10th Revision (ICD-10) criteria within 5 years before screening or positive test result(s) for alcohol and/or drugs of abuse (such as benzodiazepines, cocaines, stimulants, cannabinoids, barbiturates, opiates, phencyclidines, and tricyclic antidepressants) at screening and on Day -1

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 168 and 192 hours post-dose
  The Cmax is the maximum observed plasma concentration of rilpivirine, tenofovir, emtricitabine.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 168 and 192 hours post-dose
  The Tmax is defined as actual sampling time to reach maximum observed analyte (rilpivirine/tenofovir/emtricitabine) concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 168 and 192 hours post-dose
  The AUC (0-last) is the area under the plasma concentration-time curve for rilpivirine/tenofovir/emtricitabine from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 168 and 192 hours post-dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Elimination Rate Constant (Lambda[z]) | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 168 and 192 hours post-dose
  Lambda(z) is first-order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Elimination Half-Life (t1/2) | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 168 and 192 hours post-dose
  The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Apparent Volume of Distribution (Vdz/F) | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 168 and 192 hours post-dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vdz/F) is influenced by the fraction absorbed.
Apparent Clearance (CL/F) | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 168 and 192 hours post-dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.

SECONDARY OUTCOMES:
Number of Participants who Experience Adverse Events | Up to 17 days following study drug administration
  As a measure of safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trials, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Fukuoka, Japan

REFERENCES:
- See also: An Open-Label Study to Evaluate the Pharmacokinetics of Rilpivirine/Tenofovir/Emtricitabine After Single-Oral Administration of Rilpivirine/Tenofovir Disoproxil Fumarate/Emtricitabine Fixed-Dose Combination Tablet in Healthy Japanese Adult Male Subjects — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=10615&filename=CR107748_CSR.pdf